

## **Croydon University Hospital**

530 London Road Croydon CR7 7YE

Switchboard Tel: (020) 8401 3000

## **Informed Consent Form**

Title of Project: The effect of perineal wound infection on the anal sphincter IRAS Number: 278466

| | | IIAS Numbe | 1. 270400 | Please initial box |
|---|---|---|---|---|
| 1. | I confirm that I have read the information sheet dated (version) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | | | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | | |
| 3. | I understand that relevant sections of my medical notes and data collected during the study may be looked at by individuals from the research team, from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | | |
| 4. | I agree to my General Practitioner being informed of my participation in the study. / I agree to my General Practitioner being involved in the study, including any necessary exchange of information about me between my GP and the research team. | | | |
| 5. | I understand that photographs of my perineal wound will be taken weekly until my wound infection has resolved and wound has healed. I give permission for these photographs to be taken. | | | |
| 6. | 6. I understand that I will require an endoanal ultrasound scan weekly until my wound infection has resolved and wound healed. | | | |
| 7. | | | | |
| 8. | 8. I agree to take part in the above study. | | | |
| Name of Participant | | Date | Signature | |
| Name of Researcher taking consent | | Date | Signature | |